CLINICAL TRIAL: NCT06159452
Title: Randomized, Double-blind, Single Subcutaneous Dose, Parallel Design Study of the Tolerability of Different SAR153191 Drug Products, That Differ With Respect to Manufacturing Processes and Formulation, at Different Concentrations and Doses, in Healthy Male Subjects
Brief Title: Study of the Tolerability of Different SAR153191 Drug Products, That Differ With Respect to Manufacturing Processes and Formulation, at Different Concentrations and Doses in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TDU11373; U1111-1293-6227 (Registry Identifier: ICTRP)
Record Dates: First submitted 2023-11-28; First posted 2023-12-06 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — sarilumab

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Group A (Experimental): SAR153191 - P3 drug product concentration 1 dose 1
  Interventions: Drug: SAR153191-P3 drug product
- Group B (Experimental): SAR153191 - P2 drug product concentration 2 dose 2
  Interventions: Drug: SAR153191-P2 drug product
- Group C (Experimental): SAR153191 - P3 drug product concentration 2 dose 2
  Interventions: Drug: SAR153191-P3 drug product
- Group D (Experimental): SAR153191 - P3 drug product concentration 3 dose 3
  Interventions: Drug: SAR153191-P3 drug product
- Group B' (Experimental): SAR153191 - P2 drug product concentration 2 dose 3
  Interventions: Drug: SAR153191-P2 drug product
- Group C' (Experimental): SAR153191 - P3 drug product concentration 2 dose 3
  Interventions: Drug: SAR153191-P3 drug product
- Group E' (Active Comparator): SAR153191 - CIF3 drug product concentration 2 dose 3
  Interventions: Drug: SAR153191-C1F3 drug product

INTERVENTIONS:
Drug: SAR153191-P3 drug product — Pharmaceutical form:Solution for injection-Route of administration:Subcutaneous injection
  Other Names: SAR153191
  Arms: Group A; Group C; Group C'; Group D
Drug: SAR153191-P2 drug product — Pharmaceutical form:Solution for injection-Route of administration:Subcutaneous injection
  Other Names: SAR153191
  Arms: Group B; Group B'
Drug: SAR153191-C1F3 drug product — Pharmaceutical form:Solution for injection-Route of administration:Subcutaneous injection
  Other Names: SAR153191
  Arms: Group E'

SUMMARY:
Primary objective:

To determine the tolerability of different SAR153191 drug products that differ with respect to manufacturing processes and formulation, at different concentrations and doses, after administration of single subcutaneous doses to healthy male subjects.

Secondary objectives:

To determine the pharmacokinetic profile of the different SAR153191 drug products administered subcutaneously.

To assess the safety of the different SAR153191 drug products administered subcutaneously.

DETAILED DESCRIPTION:
Up to 35 Days

ELIGIBILITY:
Inclusion Criteria:

* Having given written informed consent prior to any procedure related to the study. Exclusion Criteria: Participants are excluded from the study if any of the following criteria apply:
* Any subject who, in the judgment of the Investigator, is likely to be noncompliant during the study, or unable to cooperate because of a language problem or poor mental development.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2010-07-09 (Actual); Primary Completion 2010-12-21 (Actual); Study Completion 2010-12-21 (Actual)

PRIMARY OUTCOMES:
Number of participants reporting injection site reactions | At predose and on Days 1, 2, 3, 4, 5, 7, 9, 11, 14, 21, and 35 following SAR153191 administration
  Injection site reactions include pain, erythema an edema.

SECONDARY OUTCOMES:
Pharmacokinetics: Cmax | At predose and on Days 1, 2, 3, 4, 5, 7, 9, 11, 14, 21 and 35 following SAR153191 administration
  Maximum plasma concentration observed
Pharmacokinetics: tmax | At predose and on Days 1, 2, 3, 4, 5, 7, 9, 11, 14, 21 and 35 following SAR153191 administration
  First time to reach Cmax
Pharmacokinetics: AUClast | At predose and on Days 1, 2, 3, 4, 5, 7, 9, 11, 14, 21 and 35 following SAR153191 administration
  Area under the plasma concentration versus time curve calculated using the trapezoidal method from time zero to the real time
Pharmacokinetics: AUC | At predose and on Days 1, 2, 3, 4, 5, 7, 9, 11, 14, 21 and 35 following SAR153191 administration
  Area under the plasma concentration versus time curve extrapolated to infinity
Pharmacokinetics: t1/2z | At predose and on Days 1, 2, 3, 4, 5, 7, 9, 11, 14, 21 and 35 following SAR153191 administration
  Terminal half-life associated with the terminal slope (λz)
Safety: Number of participants who experienced Treatment-Emergent Adverse Events (TEAEs), Treatment-Emergent Serious Adverse Events (TESAEs) and/or Treatment-Emergent Adverse Events of Special Interest (AESI) | Up to 35 Days
Incidence of anti-SAR153191 antibodies | At Day 1 predose and on Days 7, 21, and 35 (plus follow-up if positive)